CLINICAL TRIAL: NCT00410618
Title: Neurological Effects of Chemotherapy and Radiation Treatment: Colon Cancer
Brief Title: Neurological Effects of Chemotherapy and Radiation Therapy in Patients With Colon Cancer
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSCB0213; P50CA095060 (NIH); P30CA023074 (NIH); UARIZ-BSC-02-13 (Other: University of Arizona)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2012-08

CONDITIONS: Cognitive/Functional Effects; Colorectal Cancer; Long-term Effects Secondary to Cancer Therapy in Adults
Keywords: cognitive/functional effects; long-term effects secondary to cancer therapy in adults; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Mental Status and Dementia Tests; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: cognitive assessment
Procedure: magnetic resonance imaging
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Learning about the long-term effects of chemotherapy and radiation therapy on brain function may help doctors plan cancer treatments.

PURPOSE: This clinical trial is looking at the neurological effects of chemotherapy and radiation therapy in patients with colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify the nature and long-term ramifications of CNS injury as a result of cancer treatment in patients with colon cancer.

Secondary

* Analyze differences in cognitive measures and MRI data in these patients.
* Correlate MRI measures with cognitive performance in these patients.

OUTLINE: Patients undergo cognitive performance assessment and MRI.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colon cancer
* Received chemotherapy and radiotherapy for colon cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colon cancer
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2003-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Nature and long-term ramifications of CNS injury as a result of cancer treatment

SECONDARY OUTCOMES:
Differences in cognitive measures and MRI data
Relationship between MRI measures and cognitive performance

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Reminger, MD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States